CLINICAL TRIAL: NCT03786328
Title: An Outreach Collaborative Model for Early Identification and Treatment of Mental Disorder in Danish Workplaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helle Østermark Sørensen (Other)
Collaborators: Spar Nord Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Helle Østermark Sørensen, MHSc, Research Nurse, Aalborg Psychiatric Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 2013-18
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Depression, Anxiety
Keywords: Early detection and treatment
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical cases of Mental Disorder (Other): The group of individuals identified with a clinical mental disorder on the basis of the diagnostic interviews This group will be assigned to Standard Psychiatric Treatment
  Interventions: Behavioral: Standard Psychiatric Treatment
- Subclinical cases of Mental Disorder (Other): The group of individuals identified with a sub-clinical mental condition on the basis of the diagnostic interviews This group will be assigned to Preventive Psychological Treatment
  Interventions: Behavioral: Preventive Psychological Treatment

INTERVENTIONS:
Behavioral: Standard Psychiatric Treatment — Standard psychiatric treatment is offered individuals identified with a clinical mental disorder. Treatment will follow golden standard treatment in the psychiatric clinic, meaning a combination of therapy and psychopharmacological treatment.
  Arms: Clinical cases of Mental Disorder
Behavioral: Preventive Psychological Treatment — Preventive Psychological Treatment is offered individuals identified with a sub-clinical mental condition. Treatment consists of 8 sessions of cognitive-behavioural therapy.
  Arms: Subclinical cases of Mental Disorder

SUMMARY:
Depression and anxiety are prevalent mental disorders among the working population with potentially high personal and financial cost. The aim of the study is to test the applicability of an outreach collaborative model for early identification and treatment of clinical and sub-clinical mental disorders among Danish employees. applicability was examined by I) investigating the fractions of identified and treated clinical and subclinical cases, II) describing the distribution and characteristics of cases identified and III) investigating the effect of allocated treatment.

A longitudinal study design with four assessments over 16 months are applied. Six medium-large companies will be included, both public and private cooperations. Self-reporting questionnaires probing for psychopathology will be distributed to all employees in the six consecutively enrolled companies at the four time points. Employees meeting the screening criteria at T1 will be assessed diagnostically. Subjects diagnosed with a clinical mental disorder will be allocated to outpatient psychiatric treatment, and subjects with subclinical conditions will be allocated to preventive cognitive behavioural therapy. Follow-up is conducted 6 and 12 months after initiation of treatment.

Participation in the study is voluntary at all levels. Written informed consent will be obtained from participant selected for diagnostic interview and treatment.

DETAILED DESCRIPTION:
BACKGROUND:

Common mental disorders, like depression and anxiety are prevalent mental disorders among the working population with prevalence's of approximately 3% respectively. These disorder induce high personal and financial cost, due to increased number of sick days, impaired functioning - socially and professionally, reduced job satisfaction and reduced quality of life and an increased risk of loss of work.

In addition to clinical conditions, many employees are affected by symptoms of depression and anxiety at a subclinical level which can be socially inhibiting for the individual as well as negatively impacting job satisfaction, work productivity and attendance. Untreated and not early identified, these subclinical cases can lead to actual mental disorder.

In both the general population and the working population, evidence has demonstrated a high level of unmet need for mental health care and treatment. The unmet needs are partly explained by diagnostic difficulties and inadequate treatment in general practice, and partly by the fact that many individuals affected do not seek professional help.

In light of the high costs and unmet need for treatment, prevention and early detection of mental disorders among the working population ought to be a public health priority. Evidence suggests that much could be gained by investing in preventive initiatives.

Research studies within occupational mental health have mainly tested workplace-initiated stress management programmes or other universal prevention programmes using work-related outcome measures like sickness absence, work productivity and cost-effectiveness. Secondary prevention and early intervention programmes targeting mental health problems directly by using clinical standardized measures of depression or anxiety are limited, or suffer from limitations such as weak control conditions, short-term follow-up and lack of diagnostic assessment.

When targeting workplace mental health problems, it is recommended to apply a collaborative approach between workplaces and mental health specialists in order to minimize the risk of misclassification and inadequate treatment .

For this study, the investigators therefore developed an outreach secondary prevention model to be tested in collaboration between the psychiatric treatment system and workplaces in the North Denmark Region.

AIM:

The overall aim of the study was to investigate the applicability of an outreach collaborative model for early identification and treatment of clinical and sub-clinical cases of mental disorder among a Danish working population. The investigation had the following objectives:

I) To investigate the applicability of the early identification model, measured as fractions of identified clinical and subclinical cases, fraction of cases who accepted treatment and fraction of cases who completed treatment II) To describe the distribution and characteristic of clinical and subclinical cases identified by the early identification model III) To investigate the effect of allocated treatment on symptomatology for clinical and subclinical cases

METHOD:

Study design The study applies a longitudinal naturalistic design with four points of assessment (T0-T3) during a period of 16 months for each participating company. The time from T0 to T1 (4 months) constitutes a pre-treatment period and is incorporated in the design as a control period for comparison. After the second assessment (T1), screening and diagnostic assessment will be initiated. Identified cases will afterwards be allocated to treatment. Follow-up assessments are conducted after 6 months (T2) and 12 months (T3) for all employees. The assessments uses self-reporting questionnaires probing for psychopathology. All questionnaires are mailed to the employees' private postal addresses at the four points of assessment (T0-T3) followed by a reminder after two weeks in case of no response.

Participants In order to demonstrate the model's applicability in a representative sample, the investigators will enrol six medium-large companies with a minimum of 100 employees each. Companies with more than 300 employees will not be addressed due to the limitations of the available treatment capacity.

Measures The questionnaires used the Symptom Check List 90 Revised (SCL90-R) [30] as basis for identification of clinical and subclinical cases of mental disorders and follow-up to treatment. Questionnaires also collected data on demography, different work-related characteristics and job-satisfaction.

The following screening criteria for identification of clinical and subclinical cases of mental disorder is used:

i) Global Severity Index score > 0.63 or ii) values of > 0.63 in two or more subscales or iii) values of > 0.63 in the Depression subscale

Procedure Participants meeting the screening criteria at the second assessment (T1) will be invited to a diagnostic assessment in order to determine the presence of a mental disorder. The diagnostic interviews will be conducted by medical doctors at Aalborg Psychiatric Hospital, all trained and experienced user of the diagnostic instruments utilized. The presence of a mental disorder will initially be determined by use of Present State Examination (PSE). Participants assessed with a state of anxiety or depression will afterwards be rated on the Hamilton Depression Scale (HAM-D) and/or Hamilton Anxiety Scale (HAM-A) to assess the severity of the condition. Depending on the outcome of the diagnostic interview, participants will be offered two different courses of treatment:

Treatment course I: Psychiatric treatment for clinical cases Individuals diagnosed with a mental disorder according to the PSE, and with HAM-D score ≥ 18 or HAM-A score ≥ 20, will be referred to psychiatric treatment in an outpatient specialized clinic for affective disorders at Aalborg Psychiatric Hospital. The treatment will follow standard treatment procedures for psychiatric outpatients with diagnoses of depression and anxiety. Treatment is performed by trained clinicians (psychiatrists, psychologists and nurses) employed at the Clinic for Affective Disorders. The course of treatment includes medical consultations as well as psychotherapeutic sessions and treatment will continue until remission is achieved.

Treatment course II: Preventive treatment for subclinical cases Individuals assessed with subclinical conditions of depression or anxiety, defined as a HAM-D score of 13-17 or a HAM-A score of 15-19, are offered preventive treatment. This course of treatment consists of eight sessions of cognitive behavioral therapy (CBT) conducted by clinical psychologists at Aalborg Psychiatric Hospital. During the sessions, the therapeutic focus is on stress-reduction and resilience.

Statistical analysis The primary analysis are carried out by counting the number of clinical and subclinical cases identified from the early identification procedure. Secondly, the investigators will perform a descriptive analysis with the study population allocated into four groups: clinical cases, subclinical cases, untreated cases and healthy subjects. Groups will be compared at baseline (T1) on demography, work-related characteristics and the three outcome measures Global Severity Index, Depression and Anxiety.

To analyze the effect of both treatments, the investigators will use mixed effects linear regression using random intercept and with participants nested inside the companies. A p-value < 0.05 was considered statistically significant.

Ethics Information about the study are initially provided to the workplace management and the health and safety representatives and subsequently to all employees at joint open meetings.

It is emphasized that the study is voluntary at all levels. Written participant information will accompany all questionnaires. The return of the questionnaires will be considered as acceptance of participation in the questionnaire part. Written informed consent will be obtained from all participants involved in diagnostic interview and treatment. The employees are guaranteed complete anonymity in relation to their workplace and company management. The study are approved by the Danish Data Protection Agency (j. 2008-58-0028). The study was presented to the Danish Scientific Ethics Committee (N-20070016), but the need for approval was waived due to the nature of the study.

ELIGIBILITY:
Inclusion criteria:

Individuals for the diagnostic interview and treatment are selected on the basis of their response to the SCL-90-R questionnaire.

Hence, individuals are included in diagnostic interview, if scores on the SCL90-R inventory one of the following criteria:

* Global Severity Index score > 0.63 or
* values of > 0.63 in two or more subscales or
* values of > 0.63 in the Depression subscale

Exclusion criteria:

* Individuals not meeting the above screening criteria will not participate in diagnostic interview and treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Severity of Psychopathological symptoms | Measured at baseline and 6 and 12 month follow-up
  The change in severity of psychopathological symptoms are measured with the Symptom Checklist 90, revised (SCL-90-R) that is a psychiatric self-report inventory with high reliability and validity to measure overall psychological distress and to detect changes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen HO, Valentin JB, Bording MK, Larsen JI, Larsen A, Omland O. An outreach collaborative model for early identification and treatment of mental disorder in Danish workplaces. BMC Psychiatry. 2019 Jan 24;19(1):40. doi: 10.1186/s12888-019-2027-5. PMID 30678679